CLINICAL TRIAL: NCT02610114
Title: A New Method to Improve the Selection of Zygotes in the Context of Assisted Reproductive Medicine. A Randomized Controlled Blinded Monocenter Study
Brief Title: Improvement of Cell Selection in Reproductive Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jürgen Weiss (Other)
Responsible Party: Sponsor-Investigator, Jürgen Weiss, Prof. Dr. med., Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REPROLUKS 002
Record Dates: First submitted 2015-11-05; First posted 2015-11-20 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: Assisted reproductive technology (ART); zygotes; Z-score (Zygote Score); Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-Score and computer algorithm (Experimental)
  Interventions: Other: Z-Score and computer algorithm
- Z-Score (Active Comparator)
  Interventions: Other: Z-Score

INTERVENTIONS:
Other: Z-Score and computer algorithm — In addition to the routine Z-score for zygote selection, if needed, the photographs of the zygotes already taken for quality and safety reasons are analysed using the new computer algorithm. Within a few minutes it generates a score, determining the quality of the cells. The two best cells upon Z-score result and new computer algorithm result are selected for first transfer.
  Arms: Z-Score and computer algorithm
Other: Z-Score — After fertilisation pronuclei and nucleoli can be seen inside the cells by microscope. Routinely, the alignment of nucleoli can be used generating a score, the Z-score 1-4, established by Scott. Two zygotes getting the best Z-score are selected for cell culture and the cells that develop to embryo stage are used for first transfer.
  Arms: Z-Score

SUMMARY:
It is the aim of this trial to use a new computerized cell selection method, in addition to the current and world-wide used scoring system of fertilized oocytes implemented by Scott, to determine whether this leads to an increase in pregnancy rates in women undergoing assisted reproductive techniques.

DETAILED DESCRIPTION:
It is the aim of this trial to use a new computerized selection method, in addition to the current and world-wide used scoring system of fertilized oocytes (zygotes) implemented by Scott in 1998, to determine whether this leads to an increase in pregnancy rates in women undergoing assisted reproductive techniques. If successful this could in the future lead to a reduction in the numbers of embryos required to achieve a pregnancy. Transferring only one embryo means minimizing the incidence of high order multiple pregnancies.

Regularly couples gain several fertilized oocytes (zygotes) due to artificial reproductive techniques. As a routine, these cells are archived using pictures and videos for quality and safety reasons in different stages of development. Because it is planned to transfer only one or two developed embryos to the uterus, investigators have to select the zygotes with the highest potential for implantation and pregnancy. The remaining cells are preserved using vitrification.

In the study, investigators use in addition to the established Zygote-score (Z-score) by Scott a new selection method for one group of patients: The quality of the zygotes of all patients is classified according to the described Scott system. Patients are randomized to two groups. Group 1 is the control group without any further intervention. If needed for selection, the quality of the zygotes of the patients of group 2 is additionally scored with a new method. The pictures of the cells, already taken for quality and safety reasons, are taken and the cells surface is analysed using a computer algorithm.

ELIGIBILITY:
Inclusion criteria (for both male and female, couples):

* Woman with age 18 years or older
* Man with age 18 years or older
* Couples who could gain fertilized cells after In vitro fertilization (IVF) or Intracytoplasmic sperm injection (ICSI) after hormonal stimulation due to sterility treatments
* Couples presenting negative blood samples of human immunodeficiency virus (HIV) and Hepatitis B/C
* Signed routine contracts between hospital and patient wanting assisted reproductive technology (ART)
* Signed informed study consent
* Expectation of life more than 18 years
* No medical contraindication to become pregnant (female)
* Routine criteria for assisted reproductive techniques

Exclusion criteria (for female):

* Poor health status acc. to Investigator's judgement
* Expectation of life below 18 years
* Risk of ovarian hyperstimulation syndrome
* Avital cells (cells that do not further develop or die)
* Treatment due to fertility preservation, e.g. in case of cancer
* Problems after stimulation and follicle puncture
* Endometrial pathologies like polyps, submucous fibroids, etc.
* Any preceding stimulation cycle with endometrial thickness below 6mm
* Less than 4 fertilized oocytes
* Patient (and partner) wishes single embryo Transfer
* Failure to become pregnant with new zygote selection method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | min. 4 weeks after embryo transfer
  Clinical pregnancy is defined as a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.

SECONDARY OUTCOMES:
Ongoing clinical pregnancy | min. 9 weeks after embryo transfer
  Clinical pregnancy is defined as a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.
Life Birth | through study completion, an average of 40 weeks after last menstrual period
  A live birth is defined as the complete expulsion or extraction from its mother of a product of fertilization, irrespective of the duration of the pregnancy, which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation, or definite movement of voluntary muscle, irrespective of whether the umbilical cord has been cut or the placenta is attached.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Weiss, Professor, Study Chair — Luzerner Kantonsspital, Neue Frauenklinik
Locations (1):
- Neue Frauenklinik, Lucerne, Switzerland